CLINICAL TRIAL: NCT04147559
Title: Post Market Clinical Follow-Up Study for PROFEMUR® Preserve Classic Femoral Stem
Status: Enrolling by invitation | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 19H001
Record Dates: First submitted 2019-10-24; First posted 2019-11-01 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Joint Diseases
Keywords: Osteoarthritis; avascular necrosis; ankylosis; protrusio acetabuli; painful hip dysplasia
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis; Ankylosis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Total Hip Arthroplasty Implant — Single study group either newly or previously implanted with the PROFEMUR® Preserve Classic Femoral Stem combined with other Wright Medical Technology (WMT) or MicroPort Orthopedics Inc (MPO) THA components including acetabular shells, liners and femoral heads.
  Other Names: PROFEMUR® Preserve Classic Femoral Stem

SUMMARY:
Sponsor is conducting this post market clinical study to evaluate the safety and effectiveness of its PROFEMUR® Preserve Classic Femoral Stem. This type of study is required by regulatory authorities for all devices that have been approved in Europe (EU) to evaluate the medium and long-term clinical evidence. This study has been designed in accordance with MEDDEV2.12/2 (European Medical Device Vigilance System) rev2 and ISO (International Organization of Standardization) 14155:2011 guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Has previously undergone or currently has determined to undergo primary THA with the specified combination of components: PROFEMUR® Preserve Classic Stem combined with other Wright Medical Technologies (WMT) or MPO THA components including acetabular shells, acetabular liners and femoral heads.

2. Has previously undergone or currently has been determined to undergo a primary THA for any of the following:

* non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis, protrusio acetabuli, and painful hip dysplasia;
* inflammatory degenerative joint disease such as rheumatoid arthritis;
* correction of functional deformity 3. Willing and able to complete required study visits and assessments through the 10 year postoperative follow-up visit 4. Previously implanted subjects must be enrolled within 3 years of their primary THA implantation.

Exclusion Criteria:

1. Implanted with non-MPO or non-WMT components (femoral heads, acetabular shells, acetabular liners)
2. Skeletally immature (less than 21 years of age) at time of implantation
3. Has or had an overt infection at the time of implantation
4. Has or had a distant foci of infections (which may cause hematogenous spread to the implant site) at the time of implantation
5. Has or had a rapid disease progression as manifested by joint destruction or bone absorption apparent on roentgenogram at the time of implantation
6. Has or had inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable
7. Has or had neuropathic joints
8. Has or had hepatitis or HIV infection
9. Has or had a neurological or musculoskeletal disease that may adversely affect gait or weight-bearing
10. Has had a revision procedure(s) where other treatments or devices have failed; and treatment of fractures that are unmanageable using other techniques
11. Currently enrolled in another clinical investigation which could affect the endpoints of this protocol
12. Unwilling or unable to sign the Informed Consent document
13. Has documented substance abuse issue
14. Has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
15. Currently incarcerated or has impending incarceration
16. Has a medical condition, as judged by the investigator, that would interfere with the subject's ability to comply with the requirements of the protocol -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects either newly or previously implanted with the PROFEMUR® Preserve Classic Stem combined with other Wright MEdical Technology (WMT) or MPO THA components.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2033-05-01 (Estimated); Study Completion 2033-11-01 (Estimated)

PRIMARY OUTCOMES:
Component Survivorship | 10 years post-operative
  The primary objective of this study is to estimate component survivorship of the PROFEMUR® Preserve Classic Femoral Stem out to 10 years follow-up.

SECONDARY OUTCOMES:
To determine the cumulative revision rate at specified intervals out to 10 years follow-up | 10 years post-operative
  Percentage of hips that were revised or replaced at each of the intervals for Year 1, Year 3, Year 5, Year 7 and Year 10 evaluation.
Complete characterization (mean, minimum, maximum, standard deviation) of functional scores out to 10 years as assessed by HOOS. | 10 years post-operative
  The study will be reporting the final Hip Disability and Osteoarthritis Outcome Score (HOOS) which ranges from 0 to 100 with a score of 0 indicating worst hip symptoms and 100 indicating no hip symptoms.
Complete characterization (mean, minimum, maximum, standard deviation) of functional scores out to 10 years as assessed by EQ-5D-5L | 10 years post-operative
  EQ-5D-5L data will be summarized over 5 domains, namely, mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain has 5 levels: no problems, slight problem, moderate problem, severe problem, inability to perform the activity. With no problems being the best outcome and inability to perform the activity being worst outcome.
To determine proportion of subjects being satisfied and level of their satisfaction as assessed by the Forgotten Joint Score (FJS). | 10 years post-operative
  The study will be reporting forgotten joint score measures for the assessment of joint-specific patient reported outcomes. The questions focus on the patients' awareness of the implanted joint in everyday life or any unintended perception of a joint.
To determine proportion of subjects being satisfied and level of their satisfaction as assessed by the Satisfaction Survey. | 10 years post-operative
  The Satisfaction Survey consists of questions asked about how satisfied the patient is with the new implant.
To evaluate the presence of zones of radiolucencies surrounding the implanted femoral stem | 10 years post-operative
  Radiolucencies are described around 7 zones and will be reporting the number of hips with radiolucencies present at a given zone.
To characterize adverse events and adverse device effects | 10 years post-operative
  Adverse Events will be summarized as the total number of Adverse Events (AE), Adverse Device Effects (ADE) by grade, severity, and relationship to the device and surgery. Number of patients experiencing such AEs and ADEs will also be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Assini, MD, Principal Investigator — OrthoOne at Swedish Medical Center; Judd Cummings, MD, Principal Investigator — HonorHealth Research Institute
Locations (2):
- United States (2):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - HCA Research Institute, OrthoONE at Swedish Medical Center, Englewood, Colorado

IPD SHARING:
Plan to Share IPD: No